CLINICAL TRIAL: NCT04971876
Title: Prospective, Interventional, Non-Randomized, Open Label Study for the Evaluation of the Safety and Performance of an Injectable Hyaluronic Acid Filler
Brief Title: Evaluation of the Safety and Performance of an Injectable Hyaluronic Acid Filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallura Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19E2031
Record Dates: First submitted 2021-06-29; First posted 2021-07-22 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Lips Enhancement; Nasolabial Fold Correction; Midface Volume Deficit

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Lips Enhancement (Experimental): Participants treated with HLR-1 for lip enhancement, with optional Touch-Up (TU) 4 weeks afterwards
  Interventions: Device: HLR-1
- Group 2 - Nasolabial Fold Correction (Experimental): Participants treated with HLR-2 for nasolabial folds (NLFs) correction, with optional Touch-Up (TU) 4 weeks afterwards
  Interventions: Device: HLR-2
- Group 3 - Treatment of Midface Volume Deficit (Experimental): Participants treated with HLR-3 for treatment of midface volume deficit, with optional Touch-Up (TU) 4 weeks afterwards
  Interventions: Device: HLR-3

INTERVENTIONS:
Device: HLR-1 — Initial injection of HLR-1 and optional TU after 4 weeks. Maximum injection volume for each treatment session is 3mL.
  Arms: Group 1 - Lips Enhancement
Device: HLR-2 — Initial injection of HLR-2 and optional TU after 4 weeks. Maximum injection volume for each treatment session is 3mL per NLF.
  Arms: Group 2 - Nasolabial Fold Correction
Device: HLR-3 — Initial injection of HLR-3 and optional TU after 4 weeks. Maximum injection volume for each treatment session is 4mL per cheek.
  Arms: Group 3 - Treatment of Midface Volume Deficit

SUMMARY:
Evaluation of the safety and performance of the investigational device in its three concentrations for cheek and lips augmentation and correction of the nasolabial folds, assuming that the performance of the product will be demonstrated based on the responder rates observed compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subject;
* Male or female, over the age of 21;
* Seeking an aesthetic procedure on the face and can be classified into one of the following groups:

  1. Group1: Lip volume deficit with ROSSI score between 1.5 and 3 on at least the upper lip, or on both the upper and the lower lips with up to 1 point difference in ROSSI score between upper and lower lips;
  2. Group 2: Moderate to severe nasolabial folds (NLFs) with WSRS scale score 3 or 4 for each side of the face;
  3. Group 3: Mild to significant volume deficit at the cheeks level with MFVDS score 2 to 4 at each side, with up to 1 point difference in MFVDS scale score between the two sides.

     Investigator Live-Evaluator (ILE) and Injector must independently agree that the criteria is met, however concordance of the scores is not required.
* Willing to abstain from any aesthetic treatment on the face other than the treatments planned in the protocol during the study period.

Exclusion Criteria:

* Anything on the treatment site which might interfere with the evaluation (tattoo, scar, moles, too many hairs).
* Subject with mid-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease, or HIV-related disease, and/or severe malocclusion or dentofacial or maxillofacial deformities.
* Known history of multiple allergies, allergic/anaphylactic reactions including allergy to lidocaine or anaesthetics of the amide type, to hyaluronic acid products, or to Grampositive bacterial proteins.
* Inflammatory and/or infectious cutaneous disorders in or near the treatment area (herpes, acne, mycosis, papilloma, rosacea, blotches or other pathology on the treatment area, at the investigator appreciation). Subject with recurrent herpes is not eligible even if asymptomatic at time of inclusion.
* History or current autoimmune disease and/or immune deficiency.
* History of streptococcal disease (such as acute rheumatic fever or recurrent sore throats), precancerous lesions/skin malignancies, hyper- or hypo-pigmentation in face.
* Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
* Received (or is planning to receive) anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti-inflammatory drugs [oral/injectable corticosteroids or Non-Steroidal Anti-Inflammatory Drugs (NSAIDs, e.g., aspirin, ibuprofen)], or other substances known to increase coagulation time from 10 days pre- to 3 days post injection [Study device injections may be delayed as necessary to accommodate this 10-day washout period.]
* Have received at any time permanent facial implants (e.g. polyacrylamide, silicone) anywhere in the face or neck.
* Botulinum toxin injections, mesotherapy, or resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) within 6 months prior to entry in the study.
* Have received injection with a temporary bioresorbable facial dermal filler (e.g., hyaluronic acid, collagen, autologous fat, etc.) within the past 12 months prior to study start.
* Have undergone semi-permanent dermal filler treatment (e.g., calcium hydroxylapatite, poly-L-lactic acid, etc.) in the face within 24 months before enrolment.
* Have received at any time a treatment with tensor threads or gold strands on the face.
* Intensive exposure to sunlight or UV-rays within the previous month and/or foreseen during the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Responder Rate | Month 3 for Group 1, Month 6 for Groups 2 and 3
  Improvement measured by the responders rate, with a responder defined as a score improved by at least one grade from baseline, i.e. pre-treatment, as determined by the Investigator Live-Evaluator (ILE) using the relevant photo-numerical scale: ROSSI to evaluate the lip volume deficit for subjects in group 1 (scores between 1 and 5 including half scores with higher scores representing fuller lip), Wrinkle Severity Rating Scale (WSRS) for subjects in group 2 (scores between 1 and 5 where higher score represents more pronounced NLF), and Mid-Face Volume Deficit Scale (MFVDS) for subjects in group 3 (scores between 0 and 5 with lower scores representing less volume deficit).

SECONDARY OUTCOMES:
Aesthetic Improvement Based on Global Aesthetic Improvement Scale (GAIS) Subject and Investigator | Month 12
  GAIS is evaluated at Week 2 visit, Month 1, Month 3, Month 6, Month 9, Month 12
Subject's Satisfaction Based on FACE-Q | Month 12
  FACE-Q Satisfaction with Lips for Group 1, FACE-Q Appraisal of Lines: Nasolabial Folds, FACE-Q Satisfaction with Cheeks evaluated at Week 2 visit, Month 1, Month 3, Month 6, Month 9, Month 12
Performance Based on ILE Scores Compared to Baseline | Month 12
  ILE Scoring on the relevant photo-numerical scale

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (2):
  - Rosenpark Research GmbH, Darmstadt
  - Private Practice Dr.Hilton & Partner GbR, Düsseldorf
- Centrum Medyczne Evimed, Warsaw, Poland